CLINICAL TRIAL: NCT06605469
Title: Ejaculatory and Orgasmic Dysfunction Registry (Climax Registry)
Brief Title: Ejaculatory and Orgasmic Dysfunction Registry
Status: Recruiting | Type: Observational
Sponsor: Charitable Union for the Research and Education of Peyronie's Disease (Other)
Responsible Party: Sponsor
Other Study IDs: CUREPD200
Record Dates: First submitted 2024-06-13; First posted 2024-09-20 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Ejaculatory Dysfunction; Premature Ejaculation; Delayed Ejaculation; Anorgasmia; Anejaculation; Dysejaculation; Dysorgasmia
Keywords: ejaculatory dysfunction; premature ejaculation; delayed ejaculation; anorgasmia; anejaculation; dysejaculation; dysorgasmia
MeSH Terms: conditions — Ejaculatory Dysfunction; Premature Ejaculation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to evaluate the safety and efficacy of various therapies used to treat ejaculatory and/or orgasmic dysfunctions in men. The objective is to create a large, national registry designed to capture key outcomes for men being treated for ejaculatory and/or orgasmic dysfunction.

Participants will submit questionnaires about their diagnosis and treatment efficacy and multiple time intervals.

DETAILED DESCRIPTION:
The objective of the current study is to create a large, national registry designed to capture key outcomes for men being treated for ejaculatory and/or orgasmic dysfunction. To accomplish this registry, CURE PD has partnered with the Sexual Medicine Society of North America (SMSNA) to help inform sexual medicine providers of the existence of the study and to help encourage patients to enroll.

Subjects meeting criteria will be offered study entry by their local provider who will refer them to an email address to indicate their interest. Participants will then be administered questionnaires at baseline and every 3 months x 1 year, followed by every 6 months x 2 years. Patient partners will also be allowed to enroll and will receive questionnaires on the same schedule (baseline, q3 months x 1 year, q6 months x 2 years).

ELIGIBILITY:
Inclusion Criteria:

* Men being treated for either ejaculatory and/or orgasmic dysfunction
* For partners, inclusion is being a sexual partner of a man with ejaculatory and/or orgasmic dysfunction who is receiving treatment

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult men (>18) diagnosed with ejaculatory and/or orgasmic dysfunction who were recommended to begin any treatment for the condition
  For partners, inclusion is being a sexual partner of a man with ejaculatory and/or orgasmic dysfunction who is receiving treatment
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-05-30 (Actual); Primary Completion 2029-05-31 (Estimated); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
Primary Objective | 3 years
  Report subjective efficacy of therapies used to treat ejaculatory dysfunction. Study participants will have the option of indicating if they had used any treatments to treat ejaculatory disorders. If so, they will then be asked to measure its efficacy at improving their symptoms using a 1-10 scale (10 being very effective).

CONTACTS AND LOCATIONS:
Locations (1):
- The Male Fertility and Peyronie's Clinic, Orem, Utah, United States

IPD SHARING:
Plan to Share IPD: No
Deidentified data will be made available to sites which have referred patients to the registry.